CLINICAL TRIAL: NCT07309705
Title: Digital Angiography-Based Hemodynamic Assessment for Stroke Risk Stratification in Intracranial Arterial Stenosis
Brief Title: Digital Angiography-Derived Fractional Flow Assessment for Intracranial Stenosis
Acronym: CASSISS-DPR
Status: Active, not recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Suining Hospital of Traditional Chinese Medicine (Unknown); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xuanwu Jinan Hospital (Unknown); The First Affiliated Hospital of University of Science and Technology of China (Other); First Affiliated Hospital of Chongqing Medical University (Other); Jiangmen Central Hospital (Other); Hebi People's Hospital (Unknown); Shanghai Sixth People's Hospital Anhui Branch (Unknown)
Responsible Party: Sponsor
Other Study IDs: CASSISS-DPR; WKZX2025CZ0401 (Other Grant/Funding Number: Development Center for Medical Science & Technology National Health Commission of the People's Republic of China)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Atherosclerosis ICAS; Hemodynamic; Stroke
Keywords: Intracranial Atherosclerotic Stenosis; Recurrent Stroke Risk; Hemodynamic Impairment; Fractional Flow Reserve; Precision Risk Stratification
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASSISS-DPR
  Interventions: Drug: Standardized medical therapy targeting vascular risk factors and stroke prevention

INTERVENTIONS:
Drug: Standardized medical therapy targeting vascular risk factors and stroke prevention — Dual antiplatelet treatment and management of vascular risk factors, in accordance with AHA/ASA guidelines

SUMMARY:
The goal of this observational study is to learn whether a digital angiography derived fractional flow reserve (DPR) measurement can improve the prediction of stroke risk in adults with symptomatic intracranial atherosclerotic stenosis, defined as 50 to 99 percent narrowing.

The main questions it aims to answer are:

Does DPR identify patients who are at higher risk of recurrent stroke despite receiving standard medical treatment? Is DPR more accurate than traditional angiographic stenosis measurements for assessing the functional severity of intracranial arterial disease?

Participants will undergo routine digital subtraction angiography as part of their clinical evaluation. Their angiographic images will be analyzed using a computational method to estimate blood flow impairment, and they will be followed for up to 12 months to monitor stroke related outcomes.

DETAILED DESCRIPTION:
Intracranial atherosclerotic stenosis (ICAS) is a major cause of ischemic stroke, representing ~15% of cases in Western populations and up to 46.6% in Asia. Even with intensive medical therapy, annual stroke recurrence remains high (7.2-20%), prompting exploration of additional treatment strategies. Early trials such as SAMMPRIS and VISSIT suggested worse outcomes with stenting compared with aggressive medical therapy, largely due to concerns over operator experience, patient selection, and timing. Subsequent analyses showed that patients with hemodynamic compromise-such as watershed infarction and poor collaterals-have recurrence rates up to 37%, underscoring the central role of impaired cerebral perfusion.

Although more recent studies (CASSISS, BASIS) demonstrated that endovascular therapy may be safe and effective in carefully selected patients, current ICAS assessment relies primarily on stenosis severity, which correlates only weakly with true hemodynamic impairment and is insufficient for accurate risk stratification. Because symptoms arise principally from reduced perfusion, physiologic evaluation is essential.

Fractional flow reserve (FFR) is the gold standard for assessing coronary lesion significance and guiding intervention through translesional pressure gradients. Attempts to translate this approach to ICAS using invasive pressure wires have shown feasibility but remain limited by anatomical differences, lack of dedicated devices, procedural risks, and unclear outcome thresholds.

Our prior work demonstrated that intracranial translesional pressure gradients correlate strongly with cerebral blood flow in both animal models and clinical settings, validating hemodynamic relevance. To overcome the limitations of invasive measurements, the present study seeks to develop and evaluate a noninvasive, angiography-derived pressure ratio (DPR) using routine digital subtraction angiography. This method allows physiologic assessment without pressure wires and may reduce procedural risk.

The objectives of this project are to establish a computational DPR technique, determine its association with clinical outcomes, identify a hemodynamic threshold for stroke-risk stratification, and validate its performance in a prospective multicenter cohort. By enabling early identification of high-risk ICAS patients who may respond poorly to medical therapy, DPR has the potential to improve treatment selection and outcomes, ultimately advancing strategies for stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intracranial atherosclerotic stenosis (ICAS) of the anterior circulation.
2. History of an ischemic cerebrovascular event related to the target artery within the past 12 months, including ischemic stroke involving less than one-half of the middle cerebral artery territory or transient ischemic attack.
3. Age between 18 and 80 years.
4. Stenosis severity of 50% to 99% identified by transcranial Doppler ultrasound, CT angiography, or MR angiography, and confirmed as 50% to 99% stenosis on digital subtraction angiography.
5. Good compliance, willingness to sign written informed consent, and ability to complete follow-up.

Exclusion Criteria:

1. Non-atherosclerotic intracranial stenosis such as moyamoya disease, vasculitis, or arterial dissection.
2. Coexisting ipsilateral arterial stenosis greater than 50% other than the target lesion.
3. Large territorial infarction on MRI DWI involving at least one-half of the MCA territory with a modified Rankin Scale score greater than 3.
4. Contraindications to the use of antiplatelet agents or statins.
5. Inability to undergo DSA because of severe iodinated contrast allergy, severe hyperthyroidism, severe coagulation abnormalities with high bleeding risk, or severe cardiac, hepatic, or renal insufficiency.
6. Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 80 years with symptomatic intracranial atherosclerotic stenosis (50%-99%) of a major anterior-circulation artery, who experienced a target-artery-related ischemic event (ischemic stroke involving <50% MCA territory or TIA) within the past 12 months and are eligible for medical therapy and DPR evaluation.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke in the qualifying artery territory or related death within 1 year after enrollment. | Baseline to 12 months (±2 months)
  the number of participants who suffer from ischemic stroke in the qualifying artery territory or related death within 1 year after enrollment.

SECONDARY OUTCOMES:
transient ischemic attack (TIA) or ischemic stroke in the qualifying artery territory within 1 year | Baseline to 12 months (±2 months)
  the number of participants who suffer from transient ischemic attack (TIA) or ischemic stroke in the qualifying artery territory within 1 year after enrollment.
TIA related to ischemia in the qualifying artery territory within 1 year | Baseline to 12 months (±2 months)
  the number of participants who suffer from TIA related to ischemia in the qualifying artery territory within 1 year
any stroke/TIA/ death within 1 year | Baseline to 12 months (±2 months)
  the number of participants who suffer from any stroke/TIA/ death within 1 year
hemodynamic ischemic stroke in the qualifying artery territory within 1 year | Baseline to 12 months (±2 months)
  the number of participants who suffer from hemodynamic ischemic stroke in the qualifying artery territory within 1 year
embolic stroke within in the qualifying artery territory 1 year | Baseline to 12 months (±2 months)
  the number of participants who suffer from embolic stroke within in the qualifying artery territory 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Xuanwu hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: No